CLINICAL TRIAL: NCT06215625
Title: Establishment of a Feasible Smart Upper Limb Rehabilitation Model in Post-pandemic Era: Examples for Patients With Stroke and Spinal Cord Injuries
Brief Title: A Feasible Smart Upper Limb Rehabilitation Model for Patients With Stroke and Spinal Cord Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-110-563
Record Dates: First submitted 2023-12-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Spinal Cord Injuries
Keywords: stroke; spinal cord injury; robot-assisted therapy; tele-rehabilitation
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stroke: TIGER group (Experimental): Participants in the TIGER (tenodesis-induced-grip exoskeleton robot) group will operate the TIGER system. They will undergo a 30-minute home-based training program twice a day, 5 days a week for 4 weeks.
  Interventions: Other: Robot-assisted therapy
- Stroke: TOT group (Active Comparator): Participants in the TOT (task-oriented training) group will receive task-oriented training as home program. They will undergo a 30-minute home-based training program twice a day, 5 days a week for 4 weeks.
  Interventions: Other: Task-oriented training
- Spinal cord injury: TIGER group (Experimental): Participants in the TIGER (tenodesis-induced-grip exoskeleton robot) group will operate the TIGER system. They will undergo a 40-minute home-based training program once a day, 5 days a week for 4 weeks.
  Interventions: Other: Robot-assisted therapy
- Spinal cord injury: TOT group (Active Comparator): Participants in the TOT (task-oriented training) group will receive task-oriented training as home program. They will undergo a 40-minute home-based training program once a day, 5 days a week for 4 weeks.
  Interventions: Other: Task-oriented training

INTERVENTIONS:
Other: Robot-assisted therapy — The TIGER system provides assistance for activities of daily living. Continuous passive mode of TIGER system provides passive range of motion as warm-up. Functional mode TIGER system provides functional training.
  Arms: Spinal cord injury: TIGER group; Stroke: TIGER group
Other: Task-oriented training — The TOT group will practice sensorimotor techniques for warming up, and then they will practice various functional tasks based on task-oriented approach.
  Arms: Spinal cord injury: TOT group; Stroke: TOT group

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of the developed application and exoskeleton robot devices for home-based training in stroke patients and patients with spinal cord injuries. The application that uses an Internet of Things (IoT) platform to enable remote monitoring of rehabilitation progress by clinical practitioners. Simultaneously, it seeks to assist the execution of patient movements through devices.

In patients with stroke, half of the participants will be assigned to experimental group, receiving a smart upper limb motor rehabilitation system for home program. The other half will be assigned to control group, receiving a traditional home program. In patients with spinal cord injuries. Participants will follow the same allocation method for home-based intervention.

Researchers will conduct an analysis before and after intervention, examining progress in motor function, activities of daily living, and quality of life.

ELIGIBILITY:
Inclusion Criteria: For patients with stroke

* 20-79 years old.
* The score of Montreal Cognitive Assessment is more than or equal to 26.
* The unilateral hemorrhagic or ischemic participants.
* The performance of upper limb movement is affected by damage to brain cells.

Inclusion Criteria: For patients with spinal cord injury

* 20-65 years old.
* The score of Mini-Mental Status Examination is more than or equal to 25.
* Diagnosed as incomplete spinal cord injury at the C5 or C6 level.

Exclusion Criteria: For patients with stroke

* Underwent sugery on the shoulder, elbow or wrist.
* Severe pain in upper limb.
* Another muscular or neurological diseases that effects motor performance.

Exclusion Criteria: For patients with spinal cord injury

* Underwent sugery on the shoulder, elbow or wrist.
* Severe pain in upper limb.
* Another muscular or neurological diseases that effects motor performance.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity -Stroke Group - Baseline | Baseline, 4 weeks after baseline
  Fugl-Meyer Assessment - Upper Extremity is an assessment for the progress in the impairment of upper limb. 33 items in the FMA-UE include reflex activity, voluntary movement, and coordination of upper limb. 0 means movement cannot be performed, 1 means movement is partially performed and 2 means entirely performed. The minimal score is 0. The maximal score is 66. The minimal detectable change is considered 5.2.
Fugl-Meyer Assessment - Upper Extremity -Stroke Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Fugl-Meyer Assessment - Upper Extremity is an assessment for the progress in the impairment of upper limb. 33 items in the FMA-UE include reflex activity, voluntary movement, and coordination of upper limb. 0 means movement cannot be performed, 1 means movement is partially performed and 2 means entirely performed. The minimal score is 0. The maximal score is 66. The minimal detectable change is considered 5.2.
Motor Activity Log -Stroke Group - Baseline | Baseline, 4 weeks after baseline
  Motor Activity Log is a semi-structured interview to understand functional performance in individual's home. The 30 questions ask patients about perceived difficulty in daily activities, including the amount of use of their affected arm and the quality of movement. The higher scores in the former mean the higher amount of patient using his weaker arm compared to before the stroke onset. The higher scores in the latter mean the higher movement quality during daily activities. The assessment is with a range of 0 to 5. Patients can give half scores if it is more reflective for their ratings. Adding all ratings, scores will take the average. The minimal score is 0. The maximal score is 5. The minimal detectable change value is considered 1.0-1.1.
Motor Activity Log -Stroke Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Motor Activity Log is a semi-structured interview to understand functional performance in individual's home. The 30 questions ask patients about perceived difficulty in daily activities, including the amount of use of their affected arm and the quality of movement. The higher scores in the former mean the higher amount of patient using his weaker arm compared to before the stroke onset. The higher scores in the latter mean the higher movement quality during daily activities. The assessment is with a range of 0 to 5. Patients can give half scores if it is more reflective for their ratings. Adding all ratings, scores will take the average. The minimal score is 0. The maximal score is 5. The minimal detectable change value is considered 1.0-1.1.
Range of Motion -Stroke Group - Baseline | Baseline, 4 weeks after baseline
  Range of Motion is an assessment to evaluate the movements in forearm and wrist joints with a goniometer.
Range of Motion -Stroke Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Range of Motion is an assessment to evaluate the movements in forearm and wrist joints with a goniometer.
Box and Block Test -Stroke Group - Baseline | Baseline, 4 weeks after baseline
  Box and Block Test is an assessment for hand dexterity. It starts with unaffected hand and involves moving blocks one by one from a box to another one within 60 seconds. The score for each hand is calculated separately. The more blocks the patient moves in 1 minute, the better hand dexterity. The minimal detectable change value is determined for improvement in performance with 5.5 blocks or increase in 18 percent.
Box and Block Test -Stroke Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Box and Block Test is an assessment for hand dexterity. It starts with unaffected hand and involves moving blocks one by one from a box to another one within 60 seconds. The score for each hand is calculated separately. The more blocks the patient moves in 1 minute, the better hand dexterity. The minimal detectable change value is determined for improvement in performance with 5.5 blocks or increase in 18 percent.
Modified Tardieu Scale -Stroke Group - Baseline | Baseline, 4 weeks after baseline
  Modifed Tardieu Scale is an assessment for the level of spasticity at wrist joint. According to the difficulty during passive joint stretching, the score ranges from 0 to 4 in an ordinal scale. 0 means no increase in muscle tone and 4 represents unfatigable clonus occurring at a precise angle. The angle of muscle reaction is measured with a goniometer to determine where spasticity occurs during passive stretching.
Modified Tardieu Scale -Stroke Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Modifed Tardieu Scale is an assessment for the level of spasticity at wrist joint. According to the difficulty during passive joint stretching, the score ranges from 0 to 4 in an ordinal scale. 0 means no increase in muscle tone and 4 represents unfatigable clonus occurring at a precise angle. The angle of muscle reaction is measured with a goniometer to determine where spasticity occurs during passive stretching.
Semmes-Weinstein monofilament test -Stroke Group - Baseline | Baseline, 4 weeks after baseline
  Semmes-Weinstein monofilament test is an assessment for touch pressure threshold of hand. The evaluator uses nylon monofilaments of different diameters, exerting a constant force on skin for 1-1.5 seconds. The score is recorded as the finest filament that the participant could detect in at least 1 of the 3 trials. The thicker filament represents the higher score, indicating worse sensibility of hand.
Semmes-Weinstein monofilament test -Stroke Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Semmes-Weinstein monofilament test is an assessment for touch pressure threshold of hand. The evaluator uses nylon monofilaments of different diameters, exerting a constant force on skin for 1-1.5 seconds. The score is recorded as the finest filament that the participant could detect in at least 1 of the 3 trials. The thicker filament represents the higher score, indicating worse sensibility of hand.
System Usability Scale -Stroke Group - 4 weeks after baseline | 4 weeks after baseline
  System Usability Scale is a questionnaire for assessing effectiveness and satisfaction from user's subjective perspective. It consists of 10 items with a 5-point ordinal scale. 1 means strongly disagree and 5 means strongly agree. Score ranges from 0 to 100%. The threshold of good usability is 68%.
Manual Muscle Testing -Spinal Cord Injury Group - Baseline | Baseline, 4 weeks after baseline
  Manual Muscle Testing is an assessment for muscle strength in forearm and wrist muscles. It ranges from 0 to 5 in an ordinal scale. 0 means no contraction palpable and 5 means normal muscle strength.
Manual Muscle Testing -Spinal Cord Injury Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Manual Muscle Testing is an assessment for muscle strength in forearm and wrist muscles. It ranges from 0 to 5 in an ordinal scale. 0 means no contraction palpable and 5 means normal muscle strength.
Range of Motion -Spinal Cord Injury Group - Baseline | Baseline, 4 weeks after baseline
  Range of Motion is an assessment to evaluate the movements in forearm and wrist joints with a goniometer.
Range of Motion -Spinal Cord Injury Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Range of Motion is an assessment to evaluate the movements in forearm and wrist joints with a goniometer.
Functional Independence Measure -Spinal Cord Injury Group - Baseline | Baseline, 4 weeks after baseline
  Functional Independence Measure is an assessment for the functional independence status of an individual. It consists of 18 items with a 7-point ordinal scale. 1 means requiring total assistance and 7 means completely independent.
Functional Independence Measure -Spinal Cord Injury Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Functional Independence Measure is an assessment for the functional independence status of an individual. It consists of 18 items with a 7-point ordinal scale. 1 means requiring total assistance and 7 means completely independent.
Box and Block Test -Spinal Cord Injury Group - Baseline | Baseline, 4 weeks after baseline
  Box and Block Test is an assessment for hand dexterity. It starts with unaffected hand and involves moving blocks one by one from a box to another one within 60 seconds. The score for each hand is calculated separately. The more blocks the patient moves in 1 minute, the better hand dexterity. The minimal detectable change value is determined for improvement in performance with 5.5 blocks or increase in 18 percent.
Box and Block Test -Spinal Cord Injury Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  Box and Block Test is an assessment for hand dexterity. It starts with unaffected hand and involves moving blocks one by one from a box to another one within 60 seconds. The score for each hand is calculated separately. The more blocks the patient moves in 1 minute, the better hand dexterity. The minimal detectable change value is determined for improvement in performance with 5.5 blocks or increase in 18 percent.
WHO Quality of Life-BREF -Spinal Cord Injury Group - Baseline | Baseline, 4 weeks after baseline
  WHO Quality of Life-BREF is a questionnaire for assessing subjective outcome of quality of life. It consists of 26 items with a 5-point ordinal scale. 1 means very dissatisfied and 5 means very satisfied. The scores are transformed linearly to a 0-100.
WHO Quality of Life-BREF -Spinal Cord Injury Group - 4 weeks after baseline | Baseline, 4 weeks after baseline
  WHO Quality of Life-BREF is a questionnaire for assessing subjective outcome of quality of life. It consists of 26 items with a 5-point ordinal scale. 1 means very dissatisfied and 5 means very satisfied. The scores are transformed linearly to a 0-100.
Taiwanese Version of Quebec User Evaluation of Satisfaction with Assistive Technology -Spinal Cord Injury Group - 4 weeks after baseline | 4 weeks after baseline
  Taiwanese Version of Quebec User Evaluation of Satisfaction with Assistive Technology (T-QUEST) is a questionnaire for assessing user satisfaction with the use of assistive device. It consists of 12 items with a 5-point ordinal scale. 1 means not satisfied at all and 5 means very satisfied. The assessment has a range of 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chieh Kuo, Ph.D, Principal Investigator — National Cheng Kung University
Locations (2):
- Taiwan (2):
  - National Cheng-Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan